CLINICAL TRIAL: NCT05853536
Title: In Silico Trials of Surgical Interventions - Using Routinely Collected Data to Model Trial Feasibility and Design Efficiency In Vivo Randomised Controlled Trials
Brief Title: In Silico Trials of Surgical Interventions
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Leicester (Other)
Collaborators: King's College London (Other); University of Glasgow (Other); Cornell University (Other); Queen Mary University of London (Other); Newcastle University (Other); University of Bristol (Other)
Responsible Party: Sponsor
Other Study IDs: 0728UE
Record Dates: First submitted 2022-12-16; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2022-12

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard of Care: As recommended by treatment guidelines.
- Cardiovascular Intervention: Examples include:
  * Cardiac surgery - Coronary artery bypass grafting (CABG), Repair and replacement of heart valve and other cardiovascular surgery including surgery on the thoracic aorta.
  * On-pump / off-pump / minimally invasive bypass.
  * Open / Transcatheter approach for valve replacement or repair.
  * Open versus minimally invasive valve repair/ replacement.
  * Procedural coronary revascularization Percutaneous Coronary Intervention.
  * Closure of the left atrial appendage.

SUMMARY:
The project aims to establish a database of cardiovascular patients using HES and linked mortality data. This database will be used to model trials in silico with the aim of informing the design of future cardiovascular trials in the United Kingdom.

DETAILED DESCRIPTION:
Routinely collected health data such as National Health Service Hospital Episode Statistics (HES) contains a wealth of real-world longitudinal patient health data including demographics, diagnoses, procedures and other clinical information. These data can be used to address many of the existing challenges in the design and conduct of clinical trials by optimising trial design and simplifying the assessment of adherence, safety, and outcomes. When a trial concept is initiated, researchers may use HES data to explore the hypothesis and assess trial feasibility. The large-volume patient data enables a detailed understanding of the characteristics of the target patient populations and the estimation of the real-world treatment effects across different patient groups thus enabling identification of targeted populations for specific interventions. By tapping into this resource and using advanced statistical and machine learning methods, the investigators can emulate the trial and thus obtain the key trial parameters required for designing a clinical trial, minimise the number of assumptions imputed and make the design and development of clinical trials quicker, simpler, and more reliable.

ELIGIBILITY:
- The target trial protocol will be used to develop an emulated trial protocol, which will give the best approximation of the trial protocol, given the limitations and constraints of the observational data. To mimic an actual trial population, the target trial population will be matched with individual patient data from a historical trial, targeting the same population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All Adult patients (18 years and above) with cardiovascular diseases (ICD10 I00-I99) treated in NHS hospitals in England.
Sampling Method: Non-Probability Sample
Enrollment: 13977257 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) and their components | 1-Year
  As specified in the trial protocol
Major adverse cardiovascular events (MACE) and their components | 3-Year
  As specified in the trial protocol
Major adverse cardiovascular events (MACE) and their components | 5-Year
  As specified in the trial protocol

SECONDARY OUTCOMES:
Adverse Events (Arrhythmias, Dialysis, Infection, Coronary Revascularization, Reintervention) | 1-Year
  As specified in the trial protocol
Adverse Events (Arrhythmias, Dialysis, Infection, Coronary Revascularization, Reintervention) | 3-Year
  As specified in the trial protocol
Adverse Events (Arrhythmias, Dialysis, Infection, Coronary Revascularization, Reintervention) | 5-Year
  As specified in the trial protocol
Length of Hospital Stay | 1-Year
  As specified in the trial protocol
Length of Hospital Stay | 3-Year
  As specified in the trial protocol
Length of Hospital Stay | 5-Year
  As specified in the trial protocol
Rehospitalisation | 1-Year
  As specified in the trial protocol
Rehospitalisation | 3-Year
  As specified in the trial protocol
Rehospitalisation | 5-Year
  As specified in the trial protocol

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Murphy, Principal Investigator — University of Leicester
Locations (1):
- Department of Cardiovascular Sciences, University of Leicester, Clinical Sciences Wing,, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The data underlying this article were provided by National Health Service Digital under licence. Raw data may be shared with permission of National Health Service Digital.

REFERENCES:
- [Background] Pathak S, Lai FY, Miksza J, Petrie MC, Roman M, Murray S, Dearling J, Perera D, Murphy GJ. Surgical or percutaneous coronary revascularization for heart failure: an in silico model using routinely collected health data to emulate a clinical trial. Eur Heart J. 2023 Feb 1;44(5):351-364. doi: 10.1093/eurheartj/ehac670. PMID 36350978
- [Derived] Liao W, Rashid M, Brookes CL, Barber S, Turner RM, Gravel GM, Petrie MC, Lipsic E, Doenst T, Fremes S, Murphy GJ; High-Risk REVASC consortium. Study design for an emulated trial of a two arm, parallel, stratified, adaptive, RCT of CABG versus PCI in people requiring myocardial revascularisation at high risk (High-Risk REVASC). Am Heart J. 2026 Feb 2:107368. doi: 10.1016/j.ahj.2026.107368. Online ahead of print. PMID 41638385